CLINICAL TRIAL: NCT02225418
Title: Ultrasoundguided Transmuscular Quadratus Lumborum Block After Elective Laparoscopic Cholecystectomy. A Prospective, Randomized Clinical Trial.
Brief Title: Transmuscular Quadratus Lumborum Block for Laparoscopic Cholecystectomy
Acronym: TQL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of jobs
Sponsor: Jens Borglum Neimann (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor-Investigator, Jens Borglum Neimann, Associate professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBH-TQL-LC; 2013-001364-30 (EudraCT Number)
Record Dates: First submitted 2014-01-28; First posted 2014-08-26 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Cholecystitis; Pain
Keywords: Laparoscopic; Cholecystectomy; Postoperative; Pain; Quadratus lumborum; Ultrasound
MeSH Terms: conditions — Cholecystitis; Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo TQL block (Sham Comparator): 30 ml single shot TQL block with saline 0,9%
  Interventions: Drug: saline
- Active TQL block (Active Comparator): 30 ml single shot TQL block with ropivacaine 0,75%
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: naropin
  Arms: Active TQL block
Drug: saline
  Arms: Placebo TQL block

SUMMARY:
The TQL block may prove a valuable method for treating postoperative pain following scopic removal of the gall bladder.

The trial will compare active TQL block versus placebo TQL block after said operation.

The hypothesis is that active TQL block significantly will reduce postoperative pain following scopic removal of the gall bladder compared with placebo TQL block.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective laparoscopic cholecystectomy
* received oral and written information about the trial
* American Society of Anaethesiologists (ASA) classification 1-3
* NRS score > 3 upon arrival at the PACU area

Exclusion Criteria:

* Cannot cooperate
* Does not speak or understand Danish
* Allergy towards drugs used in the trial
* Large daily consumption of opioids
* Known alcohol og medicin abuse
* Difficult or impossible by ultrasound to visualise the intended nerve/tissue structures necessary to perform block
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Pain score in sitting position | 1 hour
  Numerical Rating Scale (NRS) score 1 hour after administration of TQL block

SECONDARY OUTCOMES:
Pain score at rest | 15 min, 30 min, 1 hour 2 hour 3 hour 4 hour 5 hour
  NRS score after administration of TQL block at said time points
Pain score at sitting position | 15 min 30 min 2 hour 3 hour 4 hour 5 hour
  NRS score after administration of TQL block at said time points
Total opioid consumption in PACU area | On average 3 hours
  During stay in PACU area
Opioid side effects (nausea, vomiting) | On average 3 hours
  During stay in PACU area
Length of stay in PACU area | On average 3 hours
  Total time in PACU area

CONTACTS AND LOCATIONS:
Overall Officials: Jens Børglum, MD, PhD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark